CLINICAL TRIAL: NCT06134401
Title: Effectiveness of Nebulised Hypertonic Saline to Decrease Respiratory Exacerbations in People With Neuromuscular Disease or Neurodisability: a Phase 2 Open Label Pilot Study
Brief Title: Nebulised Hypertonic Saline to Decrease Respiratory Exacerbations in Neuromuscular Disease or Neurodisability
Acronym: SPICE-UP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Pari Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23IC8597
Record Dates: First submitted 2023-11-03; First posted 2023-11-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Neuromuscular Diseases; Neurodevelopmental Disorders; Cerebral Palsy
Keywords: hypertonic saline; saline; nebulised
MeSH Terms: conditions — Neuromuscular Diseases; Neurodevelopmental Disorders; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Nebulised 6% Hypertonic saline
  Interventions: Device: saline
- Control (Placebo Comparator): Nebulised 0.9% normal saline
  Interventions: Device: saline

INTERVENTIONS:
Device: saline — nebulised

SUMMARY:
Research Aim: This study investigates whether a 12-month treatment with hypertonic saline (salty water) can reduce antibiotic use in individuals with neuromuscular disease or cerebral palsy who frequently experience chest infections due to difficulty clearing mucus from their airways.

Methodology: Participants will be randomly assigned to receive nebulised hypertonic saline (7% salt in water) or normal saline (0.9% salt in water). The study is open-label as both participants and researchers are aware of the treatment, necessary due to the differing tastes of the solutions. Two centers, Royal Brompton Hospital in London and Queens Medical Centre in Nottingham, will conduct the research.

Before starting the treatment, participants will undergo various assessments, including questionnaires to measure quality of life and treatment satisfaction, sputum/throat swab collection, lung clearance index, forced oscillation technique, electrical impedance tomography, and lung ultrasound. Once these assessments are completed, participants will take the assigned treatment at home, administered twice daily for 12 months, with monthly follow-ups regarding difficulties and chest infections. After 12 months, the treatment will cease, and participants will repeat the assessments.

Significance: This research will provide valuable insights into the efficacy of nebulised hypertonic saline for individuals with neuromuscular disease or cerebral palsy, potentially aiding both patients and doctors in making informed treatment decisions.

Dissemination: The study's findings will be shared through publication in scientific journals and presentation at conferences.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NMD or neurodisablity by a physician independent of the study, on standard criteria.
* Age 5 years and above, including adults.
* Must be able to tolerate nebulised 6% hypertonic saline.
* Must have a history of at least one respiratory exacerbation requiring antibiotic treatment with or without the need for hospitalisation in the 12 months prior to recruitment.

Exclusion Criteria:

* Patients with additional diagnosis, for example, CF, but those with aspiration and/or bronchiectasis secondary to respiratory complications of NMD will be included.
* Patients who are already prescribed daily HS in any concentration (i.e, 3%, 5%, 6%, 7%) will be excluded, but those who are on daily NS or have HS prescribed as part of their escalation plan (i.e., PRN) will be included.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Course of antibiotics for respiratory infections | from baseline to week 52
  Full courses of antibiotics as prescribed for respiratory infections, both oral and intravenous, (excluding prophylactic antibiotic prescriptions). 1 course of antibiotic would be the full treatment for one event of respiratory infection, irrespective of the number of days that the course was prescribed for.

SECONDARY OUTCOMES:
Lung clearance index | at baseline before and within 2 hours after drug response assessment, and at week 52.
  measured by multiple breath washout
Forced oscillation technique | at baseline before and within 2 hours after drug response assessment, and at week 52.
  Respiratory resistance (Rrs)
Forced oscillation technique | at baseline before and within 2 hours after drug response assessment, and at week 52.
  Respiratory reactance (Xrs).
Lung ultrasound | at baseline before and within 2 hours after drug response assessment, and at week 52.
  Global Lung ultrasound score. The global lung ultrasound score (LUS) quantifies lung aeration by translating lung ultrasound patterns into a numerical score across 12 lung regions (six areas on each side of the chest: two ventral regions, two lateral regions, and two posterolateral regions) and summing the results. The aeration pattern observed in each region is scored from 0 to 3 as follows: 0 = A pattern with ≤2 B lines; 1 = >2 separated B lines that cover ≤50% of the pleural line; 2 = B lines that cover >50% of the pleural line; or 3 = lung consolidation. In theory, the global LUS score can range from 0 (normal aeration in all regions) to 36 (severe abnormal aeration in all regions).
Electrical Impedance Tomography | at baseline before and within 2 hours after drug response assessment, and at week 52.
  Electrical impedance tomography (EIT)-based global inhomogeneity index (quantification of homogeneity of the tidal volume distribution). The image matrix in EIT consists of 32 × 32 pixels. Global inhomogeneity (GI) is calculated as the sum of the absolute differences between the median value of tidal variation and every single pixel value, divided by the sum of all impedance values, to normalise the calculated values.The smaller the GI, the more homogeneous the tidal volume is distributed within the ventilated area. A GI of zero represents a perfectly homogeneous distribution of ventilation.
Airway inflammation | baseline and at week 52
  Levels of IL-8 in sputum or throat swab.
Airway inflammation | baseline and at week 52
  Levels of IL-6 in sputum or throat swab.
Airway inflammation | baseline and at week 52
  Levels of TNF-a in sputum or throat swab.
Airway inflammation | baseline and at week 52
  Levels of IL-1b in sputum or throat swab.
Bacterial diversity | baseline and at week 52
  Operational taxonomic unit (OTU) Richness, defined as count of different species/OTUs.
Bacterial diversity | baseline and at week 52
  Pielou's eveness index. Pielou's evenness is an index that measures diversity along with species richness.
Bacterial diversity | baseline and at week 52
  Shannon diversity index. The index takes into account the number of species living in a habitat (richness) and their relative abundance (evenness).
Bacterial diversity | baseline and at week 52
  Bray-Curtis dissimilarity index. Examines the abundances of microbes that are shared between two samples, and the number of microbes found in each.
Ease of airway clearance | Once monthly for 52 weeks.
  0-10 Visual analogue scale, where 0 is most easy, and 10 is most difficult.
Health-related quality of life | At baseline and at week 51.
  Pediatric Quality of Life Inventory (PedsQL)™. 0-100 scale, where higher scores indicate better HRQOL (Health-Related Quality of Life).
Patient and main carer treatment satisfaction | weeks 12, 26, 39 and 51
  Treatment Satisfaction Questionnaire for Medication (TSQM Version 1.4). Scores range from 0 to 100, with higher scores indicating higher satisfaction.
Family impact | Baseline and at week 51.
  PedsQL™ Family Impact Module. The scale has five Likert response options, 'never', 'almost never', 'sometimes', 'often' and 'almost always' (corresponding to scores of 100, 75, 50, 25 and 0). Regarding the interpretation of the scale, higher scores indicate better functioning (less negative impact).
Health economics | baseline, week 26 and week 51.
  Quality-adjusted life years

OTHER OUTCOMES:
Recruitment rate | 1 year
  Number of participants recruited per centre per month.
Consent rate | 1 year
  Percentage of eligible participants who consented and were randomised.
Retention rate | 1 year
  Percentage of randomised participants retained with valid primary outcome data.
Adherence | 52 weeks
  Mean percentage of adherence calculated from returned ampoules count
Adherence | 52 weeks
  Pick-up rate as the percentage of picked up prescriptions from total prescribed doses
Adherence | 52 weeks
  The Medication Adherence Report Scale (MARS) Score, where each of the 5 items are summed to give a scale score ranging from 5 to 25, where higher scores indicate higher levels of reported adherence.
Compliance with monthly follow-up | 52 weeks
  Percentage of compliance with completion of monthly questionnaires.
Success rates of outcome measures | 1 year
  Percentage of participants who provided a sputum sample or throat swab
Success rates of outcome measures | 1 year
  Percentage of participants who completed acceptable measurements of Lung clearance index
Success rates of outcome measures | 1 year
  Percentage of participants who completed acceptable measurements of Forced oscillation technique
Success rates of outcome measures | 1 year
  Percentage of participants who completed acceptable measurements of Lung ulstrasound
Success rates of outcome measures | 1 year
  Percentage of participants who completed acceptable measurements of Electrical impedance tomography
Time required to complete outcome measures | 2 hours
  Time in minutes to complete acceptable measurements of Lung clearance index
Time required to complete outcome measures | 2 hours
  Time in minutes to complete acceptable measurements of forced oscillation technique
Inter-rater reliability of Lung ultrasound analysis | 1 year
  Degree of agreement among independent observers using Cohen Kappa. Cohen suggested the Kappa result be interpreted as follows: values ≤ 0 as indicating no agreement and 0.01-0.20 as none to slight, 0.21-0.40 as fair, 0.41- 0.60 as moderate, 0.61-0.80 as substantial, and 0.81-1.00 as almost perfect agreement.
Inter-rater reliability of Electrical impedance tomography analysis | 1 year
  Degree of agreement among independent observers using Cohen Kappa. Cohen suggested the Kappa result be interpreted as follows: values ≤ 0 as indicating no agreement and 0.01-0.20 as none to slight, 0.21-0.40 as fair, 0.41- 0.60 as moderate, 0.61-0.80 as substantial, and 0.81-1.00 as almost perfect agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bush, Professor, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Royal Brompton Hospital, London
  - Nottingham University Hospitals, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Data ownership rights will lie with the institution
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available after all study activities have finished. It will be available for 10 years.
Access Criteria: Data ownership rights will lie with the institution